CLINICAL TRIAL: NCT04357106
Title: COPLA Study: Treatment of Severe Forms of COronavirus Infection With Convalescent PLAsma
Acronym: COPLA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro de Hematología y Medicina Interna (Other)
Collaborators: Laboratorios Clínicos de Puebla (Laboratorios Ruiz) (Unknown)
Responsible Party: Principal Investigator, Guillermo J. RUIZ-ARGÜELLES, Dr. Guillermo J. Ruiz-Argüelles, Centro de Hematología y Medicina Interna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHMI-030420-01
Record Dates: First submitted 2020-04-14; First posted 2020-04-22 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Convalescent Plasma (Experimental): 200 ml of convalescent plasma, single dose.
  Interventions: Biological: Convalescent plasma

INTERVENTIONS:
Biological: Convalescent plasma — Convalescent plasma obtained by aphaeresis from recovered patients.

SUMMARY:
COVID-19 disease has become a very serious global health problem. Treatments for severe forms are urgently needed to lower mortality. Any procedure that improves these forms should be considered, especially those devoid of serious side effects.There is not enough published information on the use of allogeneic convalescent plasma (ACP) in the treatment of severe forms of COVID-19. The use of ACP can be combined with other treatments and has very few adverse effects. It takes 10-14 days for SARS-CoV2-infected patients to produce virus-neutralizing antibodies: within that time they can develop serious complications and die. Injecting PAC into patients with severe forms of COVID-19 shortens the period of risk while the patient produces the antibodies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with SARS-CoV2 infection who have had a serious evolution and are in an ICU
* With or without ventilatory assistance
* Treated or not with hydroxychloroquine 200 mg. every 12 hours
* Indistinct sex
* Older than 18 years
* Signed informed consent

Exclusion Criteria:

* Patients treated with the following medications: azithromycin, ritonavir / lopinavir, remdesivir, interferons, ruxolinitib, tocilizumab.
* Patients with severe kidney failure who require replacement therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-04-13 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Lung injury | 7 days
  PaO2/FiO2 relation
Overall survival | 15-30 days
  Patients survival after therapy

SECONDARY OUTCOMES:
Adverse reactions to plasma | 7 days
  Determine the incidence of side effects from plasma administration

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Hematología y Medicina Interna, Puebla City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 May 10;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub6. PMID 37162745
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 Feb 1;2(2):CD013600. doi: 10.1002/14651858.CD013600.pub5. PMID 36734509
- [Derived] Piechotta V, Iannizzi C, Chai KL, Valk SJ, Kimber C, Dorando E, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Estcourt LJ, Skoetz N. Convalescent plasma or hyperimmune immunoglobulin for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2021 May 20;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub4. PMID 34013969
- [Derived] Chai KL, Valk SJ, Piechotta V, Kimber C, Monsef I, Doree C, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Estcourt LJ, Skoetz N. Convalescent plasma or hyperimmune immunoglobulin for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2020 Oct 12;10:CD013600. doi: 10.1002/14651858.CD013600.pub3. PMID 33044747